CLINICAL TRIAL: NCT06409663
Title: A Phase 3 Open-Label, Single-Arm Study to Evaluate the Safety and Immunogenicity of a JN.1 Subvariant SARS CoV-2 rS Vaccine
Brief Title: A Strain Change Study for SARS-CoV-2 rS Vaccines
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019nCoV-315
Record Dates: First submitted 2024-05-08; First posted 2024-05-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 Infection
Keywords: coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NVX-CoV2705 vaccine (5 µg ) (Experimental): NVX-CoV2705 COVID-19 vaccine will contain rS antigen from the JN.1 subvariant of SARS-CoV-2
  Interventions: Biological: NVX-CoV2705 Vaccine

INTERVENTIONS:
Biological: NVX-CoV2705 Vaccine — All injections will be administered in a 0.5 mL injection volume at an antigenic dose of 5 µg with 50 µg Matrix-M adjuvant at each injection.
  Other Names: SARS-CoV-2 rS

SUMMARY:
The present study aims to investigate the safety and immunogenicity of the Novavax JN.1 subvariant vaccine SARS-CoV-2 rS adjuvanted with Matrix-M (NVX CoV2705) in previously vaccinated adults. A descriptive comparison will be made with participants who received the prior authorized vaccine NVX-CoV2601 in an earlier study (2019nCoV-313).

DETAILED DESCRIPTION:
This is a Phase 3, open-label, single arm study to evaluate the safety and immunogenicity of a single dose of a JN.1 subvariant severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant (r) spike (S) protein nanoparticle vaccine (SARS-CoV-2 rS) adjuvanted with Matrix-M™ (NVX CoV2705) in previously vaccinated adults.

Approximately 60 participants will be enrolled to receive a single dose of NVX CoV2705 on Day 0 and remain on study for immunogenicity until Day 28 and safety data collection up to 180 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age at time of study vaccination.
2. Previously vaccinated with ≥ 3 doses of an authorized/approved COVID-19 vaccine with the last dose administered ≥ 6 months prior to study vaccination.
3. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
4. Female participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea ≥ 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from ≥ 28 days prior to enrollment and through the end of the study.

   1. Condoms (male or female) with spermicide (if acceptable in country)
   2. Diaphragm with spermicide
   3. Cervical cap with spermicide
   4. Intrauterine device
   5. Oral or patch contraceptives
   6. Norplant®, Depo-Provera®, or other in country regulatory approved contraceptive method that is designed to protect against pregnancy
   7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle
5. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to study vaccination. Blood pressure must be ≤ 160/100 mmHg; any participant who is otherwise eligible with a blood pressure of ≥ 160/100 mmHg may be retested onsite several times over a 3-hour interval to achieve a lower blood pressure.
6. Agrees not to participate in any research involving receipt of investigational products (drug/biologic/device) including other SARS-CoV-2 prevention or treatment trials for the duration of the study.

Exclusion Criteria:

1. Current participation in research involving receipt of investigational products (drug/biologic/device).
2. Received any other vaccine within 28 days prior to study vaccination or plans to receive any other vac-cine within 28 days after study vaccination. Influenza vaccines can be administered up to 14 days before study vaccination.
3. Any known history of allergies to products contained in the investigational product in the participant's lifetime.
4. Any known history of anaphylaxis to any prior vaccine in the participant's lifetime.
5. Known history of myocarditis or pericarditis in the participant's lifetime.
6. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to study vaccination that, in the opinion of the investigator, might interfere with protocol compliance.
7. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) that requires the use of immune modulators.
8. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to study vaccination (Day 0). Persons with human immunodeficiency virus are excluded
9. Received any prohibited medication, immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to study vaccination (Day 0).
10. Active cancer (malignancy) on chemotherapy within 3 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
11. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.
12. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
13. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization [CRO], and study site personnel involved in the conduct or planning of the study).
14. Temperature of > 38°C (oral measurement) or respiratory symptoms in the past 3 days (ie, cough, sore throat, difficulty breathing) leading up to Day 0.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Incidence, duration, and severity of solicited local and systemic adverse events (AEs) | Day 7[ following 1st vaccination]
  Incidence, duration, and severity of solicited local and systemic adverse events (AEs) for 7 days following vaccination.
Incidence, severity, and relationship of any unsolicited AEs | Day 28
  Incidence, severity, and relationship of any unsolicited AEs through 28 days after vaccination.
Incidence and severity of treatment-related MAAEs, adverse events of special interest and serious adverse events interest (AESIs; predefined list, including PIMMCs, myocarditis and/or pericarditis), and serious adverse events (SAEs) | Day 180 or end of study (EoS).
  Incidence and severity of treatment-related MAAEs, adverse events of special interest and serious adverse events interest (AESIs; predefined list, including PIMMCs, myocarditis and/or pericarditis), and serious adverse events (SAEs) through day 180 or end of study (EoS).

SECONDARY OUTCOMES:
Pseudovirus neutralization titers for the JN.1 subvariant expressed as GMTs | Day 0 to Day 28
  Pseudo virus neutralization antibody responses induced by NVX CoV2705 for the JN.1 subvariant at Day 28 following study vaccination.
Pseudovirus neutralization antibody responses against the JN.1 subvariant Expressed as GMFR | Day 0 to Day 28
  Pseudovirus neutralization antibody responses of ID50 titers for the JN.1 subvariant of time points (Day 28) from Baseline
Pseudovirus neutralization antibody responses against the JN.1 subvariant Expressed as SRRs | Day 28
  Pseudovirus neutralization antibody responses of ID50 titers for the JN.1 subvariant of time points (Day 28) from Baseline
Anti-S IgG antibody responses for the JN.1 subvariant Expressed as (GMEU) | Day-0 (baseline) to Day 28.
  immunoglobulin G (IgG) antibody responses for the JN.1 subvariant at relevant time points (Days 0 and 28).
Anti-S IgG antibody responses for the JN.1 subvariant Expressed as GMFR | Frame: Day 0 and Day-28
  immunoglobulin G (IgG) antibody responses for the JN.1 subvariant at relevant time points (Days 0 and 28).
Anti-S IgG antibody responses for the JN.1 subvariant Expressed as SRRs | Frame: Day 0 and Day 28
  Immunoglobulin G (IgG) antibody responses for the JN.1 subvariant at relevant time points (Days 0 and 28).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Foothills Research Center - CCT Research, Phoenix, Arizona
  - Benchmark Research, Austin, Texas

REFERENCES:
- [Derived] Alves K, Kouassi A, Nelson J, Plested JS, Kalkeri R, Zhu M, Cloney-Clark S, Cai Z, Ahmed A, McKnight I, Mallory RM, Noriega F. Safety and immunogenicity of a single dose of a JN.1 variant COVID-19 vaccine in previously vaccinated adults: Primary analysis report of a phase 3 open-label trial. Vaccine. 2026 Feb 15;73:128164. doi: 10.1016/j.vaccine.2025.128164. Epub 2025 Dec 26. PMID 41455184